CLINICAL TRIAL: NCT02954770
Title: Fitbit® Challenge: Can we Motivate Residents to Improve Their Physical Well Being?
Brief Title: Long-term Usage of the Fitbit® Among Medical Residents
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 14-078
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Continuous Fitbit® Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fitbit® challenger: The residents who participated a Fitbit® challenge study about one year ago

SUMMARY:
This is a one year follow up survey study after a Fitbit® challenge study to determine if wearing a Fitbit® motivates residents to increase their physical activity. This study seeks to determine if residents continue to use the Fitbit® after one year.

DETAILED DESCRIPTION:
Medical training is notoriously stressful. The combination of long work hours, sleep deprivation, clinical responsibilities, and academics leaves little time for residents and fellows to consider their own health maintenance, particularly with regards to physical activity. This is problematic for both the physician and the physician's patients. Numerous studies have shown that physicians who exercise regularly and maintain normal body mass are more likely to counsel their patients on these issues. Additionally, they are more experienced in the benefits of exercise and can counsel their patients on how to incorporate exercise into a busy schedule. This is a one year follow up survey study after a Fitbit® challenge study among TriHealth residents. The purpose of the initial Fitbit® challenge study was to to determine if wearing a Fitbit® motivates residents to increase their physical activity. This study seeks to determine the long-term usage of the Fitbit®.

ELIGIBILITY:
Inclusion Criteria:

* Residents in training 18 years of age or older
* Residents who participated the initial Fitbit® challenge study

Exclusion Criteria:

* Physical impairment inhibiting the ability to walk or complete the validated questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All TriHealth residents
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Status of Fitbit® use - descriptive measure | One year after the initial Fitbit® challenge study
  This is a binary outcome, either Yes or No to survey question #20 "Do you still wear your Fitbit® originally received as part of the Fitbit® study?"

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates

IPD SHARING:
Plan to Share IPD: No